CLINICAL TRIAL: NCT06011330
Title: Efficacy , Safety, and Predictors of Fruquintinib Plus PD-1 in Refractory MSS Metastatic Colorectal Cancer in a Real-world Setting
Brief Title: Fruquintinib Plus PD-1 in Refractory MSS Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FRUPD-1
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: Fruquintinib; PD-1; pMMR/MSS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Programmed Cell Death 1 Receptor; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: fruquintinib combined with anti-PD-1 antibodies
  Interventions: Drug: Fruquintinib combined with anti-PD-1 antibodies

INTERVENTIONS:
Drug: Fruquintinib combined with anti-PD-1 antibodies — Fruquintinib (3-5mg once daily for 21 days on/7 days off) anti-PD-1 antibodies (including sintilimab, toripalimab, pembrolizumab, tislelizumab, and nivolumab).
  Other Names: programmed cell death protein 1; immune checkpoint inhibitor

SUMMARY:
The survival of the refractory CRC is dismal and therapy options are limited ，the researchers aim to investigate the efficacy, safety, and predictors of fruquintinib plus PD-1 in refractory MSS metastatic colorectal cancer in a real-world setting.

DETAILED DESCRIPTION:
The invesgators conducted a retrospective single arm, single-center study in which patients with MSS/pMMR mCRC were received fruquintinib combined with anti-PD-1 antibodies after progressed at least two lines of standard chemotherapy with or without targeted drugs such as bevacizumab and cetuximab at the Hunan Cancer Hospital from 1th January 2019 to 30th June 2022. Eligible patients were aged 18 years or older and had histologically or cytologically confirmed adenocarcinoma of the colon or rectum; with patients who have at least one non-resectable measurable lesion to evaluate by response evaluation criteria in solid tumors (RECIST version 1.1).The primary endpoint was overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. patients with MSS/pMMR mCRC who have been received Fruquintinib combined with anti-PD-1 antibodies after progressed at least two lines of standard chemotherapy with or without targeted drugs such as bevacizumab and cetuximab at the Hunan Cancer Hospital from 1th January 2019 to 30th June 2022;
2. Eligible patients were aged 18 years or older
3. had histologically or cytologically confirmed adenocarcinoma of the colon or rectum;
4. patients who have at least one non-resectable measurable lesion to evaluate by response evaluation criteria in solid tumors (RECIST version 1.1).
5. an Eastern Cooperative Oncology Group performance status of 0-2;

Exclusion Criteria:

1. Pregnancy, lactating female or possibility of becoming pregnant during the study.
2. Has not recovered from clinically relevant non-hematologic CTCAE grade ≥ 3 toxicity of previous anticancer therapy (excluding alopecia, and skin pigmentation).
3. Has symptomatic central nervous system metastases that are neurologically unstable or requiring increasing doses of steroids to control CNS disease.
4. Has severe or uncontrolled active acute or chronic infection. 5.Known carriers of HIV antibodies. 6.Confirmed uncontrolled arterial hypertension or uncontrolled or symptomatic arrhythmia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Refractory MSS Metastatic Colorectal Cancer
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | assessed up to 2 year
  Overall survival defined as the observed time from the treatment of the study until death due to any cause

SECONDARY OUTCOMES:
progress-free survival (PFS) | assessed up to 1 year
  the time from treatment initiation to the disease progression according to RECIST version 1.1 by investigator's judgement or death from any cause, whichever comes first.

OTHER OUTCOMES:
objective response rate (ORR) | assessed up to 1 year
  The ORR was calculated as the sum of the proportion of complete responses (CRs) and partial responses (PRs) according to RECIST version 1.1 criteria and using investigator's tumor assessment
disease control rate (DCR) | assessed up to 1 year
  Disease control rate has been defined as the addition of (CR + PR) rate and also stable disease (SD) rate, according to RECIST v 1.1
Treatment-Related Adverse Events (TRAE) | assessed up to 1 year
  Treatment-Related Adverse Events (TRAE) as assessed by CTCAE v5.0, including serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No